CLINICAL TRIAL: NCT00311376
Title: Safety and Efficacy Study of Botulinum Toxin Type A for the Treatment of Neurogenic Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-515
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): botulinum toxin Type A (200U)
  Interventions: Biological: botulinum toxin Type A (200U)
- 2 (Experimental): botulinum toxin Type A (300U)
  Interventions: Biological: botulinum toxin Type A (300U)
- 3 (Other): placebo; botulinum toxin Type A (200U)
  Interventions: Other: Normal Saline (Placebo); botulinum toxin Type A (200U)
- 4 (Other): placebo; botulinum toxin Type A (300U)
  Interventions: Other: Normal Saline (Placebo); botulinum toxin Type A (300U)

INTERVENTIONS:
Biological: botulinum toxin Type A (200U) — botulinum toxin Type A 200 U (tx 1) followed by botulinum toxin Type A 200 U (tx 2); injections into detrusor, at > 12 weeks interval
  Other Names: BOTOX®
  Arms: 1
Biological: botulinum toxin Type A (300U) — botulinum toxin Type A 300 U (tx 1) followed by botulinum toxin Type A 300 U (tx 2); injections into detrusor, at > 12 weeks interval
  Other Names: BOTOX®
  Arms: 2
Other: Normal Saline (Placebo); botulinum toxin Type A (200U) — Placebo (tx 1) followed by botulinum toxin Type A 200 U (tx 2); injections into detrusor, at > 12 weeks interval
  Other Names: BOTOX®
  Arms: 3
Other: Normal Saline (Placebo); botulinum toxin Type A (300U) — Placebo (tx 1) followed by botulinum toxin Type A 300 U (tx 2), injections into detrusor, at > 12 weeks interval
  Other Names: BOTOX®
  Arms: 4

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of botulinum toxin type A in treating overactive bladder in spinal cord injury or multiple sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence as a result of neurogenic overactive bladder due to spinal cord injury or multiple sclerosis
* Inadequate response to anticholinergic medication used to treat overactive bladder

Exclusion Criteria:

* History of evidence of pelvic or urologic abnormality
* Previous or current diagnosis of bladder or prostate cancer
* Urinary tract infection at time of enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2006-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (14):
- Royal Oak, Michigan, United States
- Randwick, New South Wales, Australia
- Innsbruck, Austria
- Ghent, Belgium
- Sherbrooke, Canada
- Ostrava, Czechia
- Garches, France
- Halle, Germany
- Christchurch, New Zealand
- Wroclaw, Poland
- Moscow, Russia
- Martin, Slovakia
- Lviv, Ukraine
- London, United Kingdom

REFERENCES:
- [Derived] Cuervo J, Castejon N, Khalaf KM, Waweru C, Globe D, Patrick DL. Development of the Incontinence Utility Index: estimating population-based utilities associated with urinary problems from the Incontinence Quality of Life Questionnaire and Neurogenic Module. Health Qual Life Outcomes. 2014 Oct 8;12:147. doi: 10.1186/s12955-014-0147-7. PMID 25288099
- [Derived] Chancellor MB, Patel V, Leng WW, Shenot PJ, Lam W, Globe DR, Loeb AL, Chapple CR. OnabotulinumtoxinA improves quality of life in patients with neurogenic detrusor overactivity. Neurology. 2013 Aug 27;81(9):841-8. doi: 10.1212/WNL.0b013e3182a2ca4d. Epub 2013 Jul 26. PMID 23892704
- [Derived] Ginsberg D, Gousse A, Keppenne V, Sievert KD, Thompson C, Lam W, Brin MF, Jenkins B, Haag-Molkenteller C. Phase 3 efficacy and tolerability study of onabotulinumtoxinA for urinary incontinence from neurogenic detrusor overactivity. J Urol. 2012 Jun;187(6):2131-9. doi: 10.1016/j.juro.2012.01.125. Epub 2012 Apr 12. PMID 22503020

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin Type A (300U): botulinum toxin Type A (300U)
- Botulinum Toxin Type A (200U): botulinum toxin Type A (200U)
- Placebo: Normal saline (placebo)
Period: Treatment Cycle 1
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Started | 132 | 135 | 149
Completed | 105 | 118 | 132
Not Completed | 27 | 17 | 17
Period: Treatment Cycle 2
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Started | 115 (69 from the 300U group + 46 from the Placebo group entered Cycle 2) | 125 (74 from the 200U group + 51 from the Placebo group entered Cycle 2) | 0 (Cycle 1 Placebo pts were randomized to receive 300U or 200U in Cycle 2)
Completed | 106 | 112 | 0
Not Completed | 9 | 13 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo | Total
Number analyzed (Participants) | 132 | 135 | 149 | 416
Age, Customized [Number; unit: participants]
  <40 years | 40 | 48 | 45 | 133
  Between 40 and 64 years | 83 | 73 | 95 | 251
  Between 65 and 74 years | 9 | 14 | 9 | 32
  >=75 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 80 | 76 | 245
  Male | 43 | 55 | 73 | 171

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Weekly Episodes of Urinary Incontinence
Description: Change from baseline in the weekly frequency of incontinence episodes at Week 6 after the first treatment. Incontinence is defined as involuntary loss of urine as recorded in a patient bladder diary. A negative number change from baseline indicates a reduction in incontinence episodes (improvement).
Time Frame: Baseline, Week 6
Population: Intent-to-Treat defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Number of Weekly Episodes
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Number analyzed (Participants) | 132 | 135 | 149
Number of Weekly Episodes
  Baseline | 31.1 (17.02) | 32.3 (22.76) | 28.3 (15.82)
  Week 6 | -22.7 (17.10) | -21.0 (23.77) | -8.8 (16.18)

2. Secondary Outcome: Change From Baseline in Maximum Cystometric Capacity (MCC)
Description: Change from baseline in MCC at week 6. MCC represents the maximum volume of urine the bladder holds. A positive number change from baseline represents an improvement (increase) in maximum volume of urine the bladder holds.
Time Frame: Baseline, Week 6
Population: Intent-to-Treat defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Millimeters (mL) of urine
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Number analyzed (Participants) | 132 | 135 | 149
Millimeters (mL) of urine
  Baseline | 255.8 (144.99) | 252.3 (154.37) | 256.0 (143.83)
  Week 6 | 167.7 (169.56) | 151.2 (170.59) | 15.5 (127.31)

3. Secondary Outcome: Change From Baseline in Maximum Detrusor Pressure (MDP)
Description: Change from baseline in MDP during first involuntary detrusor contraction at week 6. MDP represents the maximum pressure (peak amplitude) in the bladder during the first involuntary contraction of the bladder muscle. The greater the negative number change from baseline, the better the improvement.
Time Frame: Baseline, Week 6
Population: Intent-to-Treat defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters of water (cm H20)
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Number analyzed (Participants) | 132 | 135 | 149
Centimeters of water (cm H20)
  Baseline | 47.1 (36.30) | 51.3 (34.66) | 50.9 (38.08)
  Week 6 | -33.3 (37.75) | -35.1 (35.67) | -2.4 (43.41)

4. Secondary Outcome: Change From Baseline in Total Score on Incontinence Quality of Life (I-QOL) Questionnaire
Description: Change from baseline in I-QOL questionnaire total score at Week 6, as completed by the patient. The I-QOL is a validated, disease-specific quality of life (QOL) questionnaire containing 22 questions designed to measure impact of urinary incontinence on patients' lives. Each question is answered on a 5-point scale (1 = worst QOL and 5 = best QOL). The scores are totaled over the 22 questions and normalized to a score of 0-100 (0 = worst QOL and 100= best QOL). A positive change from baseline represents an improvement
Time Frame: Baseline, Week 6
Population: Intent-to-Treat defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Number on a Scale (Score)
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Number analyzed (Participants) | 132 | 135 | 149
Number on a Scale (Score)
  Baseline | 32.18 (18.609) | 33.95 (18.021) | 35.06 (18.066)
  Week 6 | 32.92 (23.849) | 26.90 (26.813) | 10.81 (18.413)

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were randomized AND treated. S(AE)s are displayed for the placebo-controlled treatment Cycle 1.
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Serious Adverse Events (participants affected / at risk) | 30/127 | 24/135 | 22/145
Other Adverse Events (participants affected / at risk) | 82/127 | 92/135 | 70/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (300U) (N=127) | Botulinum Toxin Type A (200U) (N=135) | Placebo (N=145)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Adverse Drug Reaction (General disorders) | 1 | 0 | 0 — Event not related to study drug, but to concomitant medication
Death (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0 — Event related to central intravenous catheter
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0
Central nervous system abscess (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Eschar (Injury, poisoning and procedural complications) | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 10 | 0 | 3
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 — Event not related to study medication; related to underlying adverse event of urinary tract infection
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Botulinum Toxin Type A (300U) (N=127) | Botulinum Toxin Type A (200U) (N=135) | Placebo (N=145)
Nausea (Gastrointestinal disorders) | 8 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 8 | 4
Pyrexia (General disorders) | 4 | 10 | 5
Fatigue (General disorders) | 4 | 8 | 6
Urinary tract infection (Infections and infestations) | 64 | 66 | 49
Vulvovaginal mycotic infection (Infections and infestations) | 3/89 | 6/80 | 2/76 — Percentages for this adverse event were calculated based on the number of female patients in each group
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 4 | 4
Multiple sclerosis relapse (Nervous system disorders) | 12 | 1 | 3
Headache (Nervous system disorders) | 7 | 4 | 4
Urinary retention (Renal and urinary disorders) | 22 | 27 | 5
Bladder pain (Renal and urinary disorders) | 7 | 2 | 2
Haematuria (Renal and urinary disorders) | 6 | 7 | 4
Hypertension (Vascular disorders) | 7 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.